CLINICAL TRIAL: NCT02184546
Title: Outcomes Data of Adipose Stem Cells to Treat Parkinson's Disease
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: StemGenex (Industry)
Responsible Party: Sponsor
Other Study IDs: SVF01PD; ASCPD-01
Record Dates: First submitted 2014-07-03; First posted 2014-07-09 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The purpose of this study is to determine the impact that treatment with a cellular concentrate derived from an individual's own fat, known as the stromal vascular fraction (SVF), has on the quality of life of people with Parkinson's disease (PD). SVF contains components with "regenerative" properties, including stem cells that may be capable of ameliorating specific disease conditions. This study is designed to evaluate quality of life changes in individuals with PD for up to 12 months following SVF treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects scheduled for a stem cell/SVF treatment
* Subjects diagnosed with idiopathic Parkinson's disease
* Subjects ages 18 years and older
* Subjects willing and able to sign informed consent
* Subjects willing and able to perform follow up interviews and surveys

Exclusion Criteria:

* Subjects with additional major health diagnoses
* Subjects that are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community Sample
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2014-07; Primary Completion 2019-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Overall Quality of Life Over the Course of a 12 Month Period as Measured by the Parkinson's Disease Quality of Life Questionnaire (PDQUALIF) | Baseline, 12 months
  The change from baseline over the course of 12 months using participants' assessment of their overall quality of life. Mean scores will be used for baseline (day 0) and all interviews up to month 12 (months 1, 3, 6, and 12). Answer options are graded according to one of seven various five-point Likert response scales.

SECONDARY OUTCOMES:
Change from Baseline in Social and Role Function at Month 12 as Measured by Participants Using the Parkinson's Disease Quality of Life Questionnaire (PDQUALIF) The Social and Role Function Subscale | Baseline, Month 12
  Participant assessment of the change in their social functioning from baseline to month 12 using the PDQUALIF social and role function subscale
Change from Baseline in Self Image and Sexuality at Month 12 as Measured by Participants Using the Parkinson's Disease Quality of Life Questionnaire (PDQUALIF) The Self Image and Sexuality Subscale | Baseline, Month 12
  Participant assessment of the change in their self image and sexual functioning from baseline to month 12 using the PDQUALIF self image and sexuality subscale
Change from Baseline in Sleep at Month 12 as Measured by Participants Using the Parkinson's Disease Quality of Life Questionnaire (PDQUALIF) The Sleep Subscale | Baseline, Month 12
  Participant assessment of the change in their sleep quality from baseline to month 12 using the PDQUALIF sleep subscale
Change from Baseline in Outlook at Month 12 as Measured by Participants Using the Parkinson's Disease Quality of Life Questionnaire (PDQUALIF) The Outlook Subscale | Baseline, Month 12
  Participant assessment of the change in their life outlook from baseline to month 12 using the PDQUALIF outlook subscale
Change from Baseline in Physical Functioning at Month 12 as Measured by Participants Using the Parkinson's Disease Quality of Life Questionnaire (PDQUALIF) The Physical Functioning Subscale | Baseline, Month 12
  Participant assessment of the change in their physical functioning from baseline to month 12 using the PDQUALIF physical functioning subscale
Change from Baseline in Independence at Month 12 as Measured by Participants Using the Parkinson's Disease Quality of Life Questionnaire (PDQUALIF) The Independence Subscale | Baseline, Month 12
  Participant assessment of the change in their feeling of independence from baseline to month 12 using the PDQUALIF independence subscale
Change from Baseline in Urinary Function at Month 12 as Measured by Participants Using the Parkinson's Disease Quality of Life Questionnaire (PDQUALIF) The Urinary Function Subscale | Baseline, Month 12
  Participant assessment of the change in their urinary function from baseline to month 12 using the PDQUALIF urinary function subscale
Change from Baseline in Global Health-Related Quality of Life at Month 12 as Measured by Participants Using the Parkinson's Disease Quality of Life Questionnaire (PDQUALIF) The Global HRQoL Subscale | Baseline, Month 12
  Participant assessment of the change in their overall health-related quality of life from baseline to month 12 using the PDQUALIF global HRQoL subscale

CONTACTS AND LOCATIONS:
Locations (1):
- StemGenex, San Diego, California, United States